CLINICAL TRIAL: NCT04570007
Title: Vitreous Fragments Length After Pars Plana Vitrectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale Policlinico San Martino (Other)
Responsible Party: Sponsor
Other Study IDs: 2/2020
Record Dates: First submitted 2020-09-24; First posted 2020-09-30 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-09

CONDITIONS: Vitreous Disorder; Vitreous Anomalies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — vitreous collagen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Pars Plana Vitrectomy — removal of vitreous with vitreous cutter

SUMMARY:
To measure vitreous collagen fragments length after pars plana vitrectomy performed at different cut rates

DETAILED DESCRIPTION:
Pars plana vitrectomy consists in the removal of vitreous obtained with a vitreous cutter. The instruments attracts vitreous in its port through active suction and cuts with a blade at different cut rates. There is no consensus as to which cut rate would be ideal in order to minimize traction, neither there is agreement on whether increasing cut rates generate shorter collagen fragments or the fluid turbulence creates unpredictable flows at the port generating fragments of different length.

The investigators plan to gather vitreous cut at 1,000, 2,000, 4,000, 8,000 and 16,000 cuts per minute and measure vitreous collagen average length

ELIGIBILITY:
Inclusion Criteria:

* patient undergoing pars plana vitrectomy for:
* macular pucker
* macular hole-
* retinal detachment
* age >18

Exclusion Criteria:

* unwilling to participate
* previous trauma
* vitreous haemorrhage

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients over 18 undergoing pars plana vitrectomy for macular surgery or retinal detachment
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2020-09-20 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-12-10 (Estimated)

PRIMARY OUTCOMES:
collagen fragment molecular weigth | at time of surgery
  collagen passed through the vitreous cutter is examined with regard to collagen moecular weigth

CONTACTS AND LOCATIONS:
Overall Officials: Tommaso Rossi, Principal Investigator — IRCCS Policlinico San MArtino
Locations (1):
- IRCCS Policlinico San Martino, Genova, RM, Italy

IPD SHARING:
Plan to Share IPD: No